CLINICAL TRIAL: NCT05025943
Title: Omega-3 Fatty Acid Dietary Intervention for Dyslipidemia of Obesity in Children 10 to <18 Years of Age: O3DI Study
Brief Title: Omega-3 Fatty Acid Dietary Intervention (O3DI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O3DI
Record Dates: First submitted 2021-08-16; First posted 2021-08-30 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard lifestyle intervention + omega-3 fatty acid enriched diet (Experimental): American Heart Association Target Diet/Standard Lifestyle Intervention (SLI) + omega-3 fatty acid enriched foods
  Interventions: Other: Diet intervention
- Standard lifestyle intervention (Active Comparator): American Heart Association Target Diet/Standard Lifestyle Intervention (SLI)
  Interventions: Other: Control group

INTERVENTIONS:
Other: Diet intervention — The intervention group will receive diet counseling and information to implement a standard lifestyle intervention plus omega-3 fatty acid enriched foods Diet assessment and counseling provided throughout study.
  Other Names: Standard lifestyle intervention + omega-3 fatty acid enriched diet
  Arms: Standard lifestyle intervention + omega-3 fatty acid enriched diet
Other: Control group — The control group will receive diet counseling and information to implement a standard lifestyle intervention Diet assessment and counseling provided throughout study.
  Other Names: Standard lifestyle intervention
  Arms: Standard lifestyle intervention

SUMMARY:
Elevated cholesterol, including triglyceride levels, can lead to the development of cardiovascular disease in adulthood. A diet that is rich in omega-3 fatty acids (O3FA) can improve triglyceride levels in a way that is safe and does not require medication.

This is a single-center, prospective, unblinded, randomized-controlled dietary intervention study to assess the impact of an omega-3 fatty acid diet compared to a standard lifestyle intervention on serum triglyceride in patients with hypertriglyceridemia. The study consists of an 8-week dietary treatment period followed by an 8-week observation period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients who are 10 -17 years of age
2. BMI greater than or equal to the 85th percentile
3. Clinical serum triglyceride level >150 mg/dl and < 500 mg/dl performed between 3 months and 1 week prior to study visit 1
4. Ability to follow the study procedures and adhere to the diet counseling recommendations
5. Written parental permission and assent are obtained prior to any research procedures

Exclusion Criteria:

1. Type 2 DM (hemoglobin A1C >6.6%)
2. Isotretinoin use
3. Chronic kidney disease (CKD)
4. Uncontrolled hypothyroidism
5. Warfarin use
6. Liver disease (NAFLD is allowed)
7. Renal disease
8. Corticosteroid use
9. Omega-3 fatty acid use (prescription or supplement)
10. Allergy to fish and/or nuts
11. Currently pregnant or planning to become pregnant during the course of this trial - confirmed by date of LMP/querying family
12. Any significant medical condition which the investigator believes would interfere with participation in this study

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
change in serum triglyceride level after an 8-week diet intervention compared to baseline | 8 weeks
  The study will test whether omega-3 fatty acid enriched diet is associated with a 20% or greater reduction in serum triglyceride levels.

SECONDARY OUTCOMES:
change red blood cell omega-3 fatty acid content / index after an 8-week diet intervention compared to baseline | 8 weeks
  Total levels of omega-3 fatty acids in red blood cell membrane phospholipids are measured. Percentages are reported as an index. The study will identify the index/total omega-3 fatty acid in red blood cells following initiation of an omega-3 fatty acid enriched diet.

CONTACTS AND LOCATIONS:
Overall Officials: Carissa Baker-Smith, MD, MPH, MS, Principal Investigator — Nemours Cardiac Center, Nemours Children's Hospital Delaware
Locations (1):
- Nemours Cardiac Center, Nemours Children's Hospital Delaware, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No